CLINICAL TRIAL: NCT06655896
Title: A Phase II, Multi-part, Randomized, Open-label, Assessor-blinded, Active-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Rapcabtagene Autoleucel Versus Rituximab Treatment in Participants With Severe Refractory Diffuse Cutaneous Systemic Sclerosis
Brief Title: Phase 2 Study Evaluating Rapcabtagene Autoleucel in Participants With Diffuse Cutaneous Systemic Sclerosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CYTB323K12201; 2023-510380-34-00 (Other: CTIS number)
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Scleroderma, Diffuse
Keywords: Diffuse cutaneous systemic sclerosis (dcSSc); Scleroderma, Diffuse; revised Composite Response Index in Systemic Sclerosis (rCRISS); modified Rodnan skin score (mRSS); forced vital capacity (FVC)
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Rituximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study investigator and the participant will be unblinded to the study treatment. A blinded assessor will perform the efficacy assessments to minimize bias in data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rapcabtagene autoleucel arm (Experimental): rapcabtagene autoleucel
  Interventions: Biological: rapcabtagene autoleucel
- rituximab arm (Active Comparator): rituximab
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rapcabtagene autoleucel — single infusion of rapcabtagene autoleucel
  Arms: rapcabtagene autoleucel arm
Biological: rituximab — rituximab intravenous infusion (i.v.) as per protocol
  Arms: rituximab arm

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of rapcabtagene autoleucel (administered once following lymphodepletion) in participants with severe refractory diffuse cutaneous systemic sclerosis relative to rituximab.

DETAILED DESCRIPTION:
This is a phase 2, multi-part, five-year, randomized, open-label, assessor-blinded, multicenter study to evaluate the efficacy and safety of rapcabtagene autoleucel versus rituximab in participants with severe refractory diffuse cutaneous systemic sclerosis (dcSSc). This study comprises two cohorts:

* A Lead-in Cohort enrolling participants to receive rapcabtagene autoleucel.
* A Randomized Cohort enrolling participants to receive rapcabtagene autoleucel or rituximab. Participants in the rituximab arm whose disease is not fully controlled may receive rapcabtagene autoleucel treatment once the participant is confirmed to be eligible per protocol.

After end of study, participants who received rapcabtagene autoleucel infusion will enter a long-term follow-up (LTFU) period after rapcabtagene autoleucel infusion. This LTFU will be described in a separate study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must fulfill the 2013 American College of Rheumatology/ European League Against Rheumatism classification criteria for systemic sclerosis and meet the diffuse cutaneous SSc (dcSSc) subset classification according to LeRoy.
2. Disease onset from the first non-Raynaud symptoms attributable to SSc (e.g., puffy hands, scleroderma, digital ulcers, arthralgia, dyspnea) within 7 years prior to the Screening visit.
3. Severe, progressive systemic sclerosis disease defined by at least one of the following:

   * Progressive systemic sclerosis-associated interstitial lung disease
   * Severe, progressive systemic sclerosis skin disease
   * Clinically significant systemic sclerosis-associated cardiac involvement at Screening
4. All recommended vaccinations received according to institutional, local or global guidelines for immuno-compromised patients.

Exclusion Criteria:

1. Any condition during Screening that could prevent a complete washout of medications as required per protocol or could otherwise make the participant ineligible for anti-CD19 CAR-T therapy and further participation in the study, as judged by the Investigator.
2. Participants with history of hypersensitivity to excipients in rapcabtagene autoleucel or to rituximab.
3. Any participant for whom treatment with rituximab is clinically inappropriate in the opinion of the investigator.
4. Any medical conditions that are not related to SSc that, in the opinion of the Investigator, would jeopardize the ability of the participant to tolerate lymphodepletion and anti-CD19 CAR-T cell therapy.
5. Rheumatic disease other than dcSSc, (except secondary Sjogren's syndrome or scleroderma myopathy),including limited cutaneous systemic sclerosis (lcSSc) or sine scleroderma at Screening.
6. Participants with pre-existing pulmonary hypertension.
7. Significant renal pathology at Screening.
8. Participants with uncontrolled stage II hypertension at Screening.
9. Vaccination with live attenuated vaccines within 6 weeks prior to randomization.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2032-08-30 (Estimated)

PRIMARY OUTCOMES:
Achievement of a treatment response as per the Revised Composite Response Index in Systemic Sclerosis 50 (rCRISS50) definition at Week 52. | Week 52
  To demonstrate the superiority of rapcabtagene autoleucel as a single infusion compared to rituximab, with respect to the proportion of participants achieving a Revised Composite Response Index in Systemic Sclerosis 50 (rCRISS50) response at Week 52.
  This response is assessed across 5 assessment domains: (1) modified Rodnan Skin Score (mRSS), (2) Health Assessment Questionnaire Disability Index (HAQ-DI), (3) patient global assessment (PGA), (4) physician global assessment (PhGA) and (5) percent-predicted forced vital capacity (FVC%).

SECONDARY OUTCOMES:
Change from baseline in Forced Vital Capacity (FVC)% predicted at Week 52 | Baseline, Week 52
  Change from baseline in FVC % predicted
Change from baseline in modified Rodnan Skin Score (mRSS) at Week 52. | Baseline, Week 52
  The modified Rodnan Skin Score (mRSS) is a clinical tool used to assess skin thickness in patients with systemic sclerosis (scleroderma). It involves palpating the skin and rating its thickness on a scale from 0 to 3 across 17 different body sites. The total score is the sum of the individual scores from all 17 sites, ranging from 0 (normal) to 51 (severe).
Change from baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 52. | Baseline, Week 52
  The Health Assessment Questionnaire Disability Index (HAQ-DI) is a widely used tool to measure a patient's level of functional ability and disability. It consists of 20 questions that cover eight domains of daily living activities: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Each question is rated on a scale from 0 (without difficulty) to 3 (unable to do).
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to end of study, assessed up to approximately 5 years
  The distribution of adverse events will be done via the analysis of frequencies for Adverse Event (AEs) and Serious Adverse Event (SAEs) through the monitoring of relevant clinical and laboratory safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (76):
- United States (13):
  - UCLA, Los Angeles, California
  - UCSF, San Francisco, California
  - Sutter Health Network, San Pablo, California
  - FL Medical Clinic Orlando Health, Zephyrhills, Florida
  - Northwestern University, Chicago, Illinois
  - University Of Iowa, Iowa City, Iowa
  - Boston Medical Center, Boston, Massachusetts
  - Michigan Med University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - James Cancer Hospital, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Avera Cancer, Sioux Falls, South Dakota
  - LDS Hospital, Salt Lake City, Utah
- Australia (2):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Darlinghurst, New South Wales
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, São Paulo, São Paulo, Brazil
- Czechia (2):
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Aarhus N, Denmark
- France (7):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
- Germany (9):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Ulm
- Hungary (2):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (11):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Udine, UD
- Japan (7):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kyoto
- Novartis Investigative Site, Utrecht, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (9):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Valencia
- Switzerland (3):
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.